CLINICAL TRIAL: NCT06823830
Title: Clinical、metabolomics and the Study of Intestinal Flora of Jinfeng Pills in the Treatment of Polycystic Ovary Syndrome
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: JFPILL202306
Record Dates: First submitted 2023-07-11; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-07

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Jinfeng Pill Group (Experimental)
  Interventions: Drug: Jinfeng Pill
- Jinfeng pill+Diane-35 Group (Experimental)
  Interventions: Drug: Jinfeng Pill
- Jinfeng Pill(placebo)+Diane-35 Group (Active Comparator)
  Interventions: Drug: Jinfeng Pill

INTERVENTIONS:
Drug: Jinfeng Pill — Jinfeng pills were compared with Diane-35 group and Jinfeng pills combined with Diane-35 group were compared with Diane-35 alone.

SUMMARY:
The goal of this clinical trial is to compare the clinical effect of Jinfeng Pill and Diane-35 in patients with PCOS. The main questions it aims to answer are: a. Comparison of the efficacy of the drugs separately and in combination. To explore the possible mechanism of Jinfeng pills. Participants will be treated for three months with monthly follow-up. Blood and stool samples should be collected.

DETAILED DESCRIPTION:
In this study, the clinical efficacy of Jinfeng pill in the treatment of PCOS was evaluated, and the clinical systems biology research system was introduced to discuss the clinical mechanism of Jinfeng pill in the treatment of PCOS from the perspectives of metabolomics and intestinal flora, etc., and an integrated biomarker index system was established to evaluate the efficacy of Jinfeng pill in the treatment of PCOS. To clarify the action mechanism and pharmacodynamic material basis of Jinfeng pills in treating PCOS. According to the previous study, a total of 105 participants were included. They were required to complete three months of treatment and monthly follow-up visits. The main therapeutic index was improved level of sex hormone. Secondary efficacy indexes included symptom scale score and TCM scale score. It has also been explored to incorporate changes such as metabolomic molecules and gut microbiota.

ELIGIBILITY:
Inclusion Criteria:

1. Meet the diagnostic criteria for PCOS: refer to the 2003 Rotterdam standard.
2. In the past 1 month, no relevant drugs or surgery were used, including periodic use of progesterone, short-acting compound oral contraceptives, sequential treatment of estrogen progesterone, spironolactone, pioglitazone, acarboxylose, and related Chinese medicine.
3. Subjects (or their legal representatives) must understand the nature of the study and sign informed consent.
4. Patients with other chronic diseases under stable control should maintain the original treatment regimen during the study period.

Exclusion Criteria:

1. Patients with other endocrine diseases, such as adrenal cortical hyperplasia or tumor, Cushing's syndrome, thyroid disease, hyperprolactinemia, androgen secreting tumors, etc.;
2. Patients who have used related drugs in the past 1 month, including sex hormone drugs, insulin sensitizers, including metformin, liraglutide and other drugs;
3. Substance abuse or dependence (alcohol or drugs) within the past 3 months; Heavy smokers (smokers who smoke 20 or more cigarettes a day);
4. Patients with serious or unstable physical diseases, including liver, kidney, gastrointestinal, cardiovascular, respiratory, endocrine, neurological, immune or blood system diseases, mental disorders;
5. Lactating or pregnant women, or women within 1 year after childbirth;
6. Previous allergy to the experimental drug;
7. History of thromboembolic disease or tendency to thrombosis;
8. Participated in a clinical trial of another investigational drug within 1 month prior to inclusion in this study (first interview);
9. Those who meet the inclusion criteria, do not follow medical advice, cannot judge the efficacy or have incomplete data to evaluate the efficacy.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 105 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-02-28 (Estimated); Study Completion 2025-02-28 (Estimated)

PRIMARY OUTCOMES:
Sex hormone | twice (before and after 3-month treatment)
  FSH、 LH、 E2、 T、 PRL、 DS、 AMH

SECONDARY OUTCOMES:
Menstrual status | everyday during 3-month treatment
  patients were asked to record the day they menstruating, menstruation duration and the flow level (light/ medium/ heavy) and concomitant symptom
acne score | twice (before and after 3-month treatment)
  applying Global Acne Grading System（GAGS）, scored by gynecologist
hirsutism score | twice (before and after 3-month treatment)
  applying Ferriman-Gallwey scoring system, scored by gynecologist
Traditional Chinese Medicine Symptom Score | every month during 3-month treatment
  patient self-assessment scale, in Chinese
36-Item Short Form Survey | every month during 3-month treatment
  SF-36 is a self-reported survey that assesses physical and mental health outcomes.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No